CLINICAL TRIAL: NCT02579161
Title: Trial of Randomized Antibiotic Administration in Percutaneous Nephrolithotomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 14-003
Record Dates: First submitted 2014-06-19; First posted 2015-10-19 (Estimated); Results first posted 2023-03-14 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Kidney Stones
Keywords: Percutaneous Nephrolithotomy; Kidney Stones; Antibiotics
MeSH Terms: conditions — Kidney Calculi | interventions — Cephalosporins; Cefazolin; Fluoroquinolones; Ciprofloxacin; Clindamycin; Lincosamides; Ampicillin; Gentamicins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Antibiotics for a 24 hour period (Active Comparator): Antibiotics for a 24 hour period
  Intervention drug to be determined based on patient history etc.
  Interventions: Drug: cephalosporins; Drug: Fluoroquinolones; Drug: Clindamycin; Drug: Ampicillin/Gentamicin
- Continued antibiotics (Active Comparator): Continued antibiotics until the removal of any external catheters
  Intervention drug to be determined based on patient history etc.
  Interventions: Drug: cephalosporins; Drug: Fluoroquinolones; Drug: Clindamycin; Drug: Ampicillin/Gentamicin

INTERVENTIONS:
Drug: cephalosporins — Patients were randomly assigned to the interventional arm or the control arm through stratified randomization. In addition to perioperative antibiotics, those in the interventional arm only received antibiotic course for up to 24 hours after procedure, while those in the control arm received antibiotics until external catheters were removed based on surgeon preference. Ancef, a 1st generation cephalosporin, was used as the primary antibiotic, which was started within 60 minutes of the procedure. Dosing was 1 gram IV every 8 hours and was adjusted for renal dosing as needed
  Other Names: ancef
Drug: Fluoroquinolones — If the patient has an allergy to penicillin or cephalosporin, then Ciprofloxacin was used instead and started within 120 minutes of the procedure at 400mg IV and would be continued every 12hrs if patient has a normal creatinine clearance
  Other Names: ciprofloxacin
Drug: Clindamycin — If allergic to penicillin, cephalosporins, and fluoroquinolones, 900 mg Clindamycin started within 60 minutes prior to initial surgical incision.
  Other Names: Lincosamides
Drug: Ampicillin/Gentamicin — 5 mg/kg as a single dose of Gentamicin within 60 minutes prior to surgical incision; given in combination with 2 grams of ampicillin in cases where allergic to fluoroquinolone and cephalosporin
  Other Names: Penicillinase-sensitive penicillin\Aminoglycoside

SUMMARY:
The Investigators objective is to compare the clinical efficacy of a single-day protocol with a short-course protocol for PCNL. The investigator hope is to reduce the use of possibly unnecessary prolonged antibiotic use, reduce hospital costs and prevent the further propagation of resistant microbes.

DETAILED DESCRIPTION:
For large renal stone burdens and/or complex stones, Percutaneous Nephrolithotomy (PCNL) has become the mainstay for treatment, replacing open kidney stone surgery since it's introduction in 1976. However, PCNL is not without its complications, specifically infectious. The procedure carries up to 25% incidence of infectious complications with approximately 1% rate of severe sepsis even with completely sterile conditions. Therefore, the use of antibiotics becomes paramount, but to date there are no PNCL specific guidelines for the appropriate duration and class of antibiotics. This fact leaves the practicing urologists to their own subjective experiences to the guide them. In addition, in an age where there are increasing numbers of resistant microbes the judicious use of antibiotics is in even more paramount.

The investigators of this project, purpose a randomized intention to treat prospective study to explore the duration and type of antibiotics in a larger population then previously studied. The investigators hypothesize that there will be no difference in complications between two groups: 1) 24 hours of perioperative antibiotics versus 2) Continued antibiotics until the removal of any external catheters. The investigators will model the antibiotics choices and duration after the 2013 American Urological Association, (AUA) Urologic Surgery Antimicrobial Prophylaxis recommendations, modified by our local antibiogram as necessary. The investigators' objective is to compare the clinical efficacy of a single-day protocol with a short-course protocol for PCNL. Our hope is to reduce the use of possibly unnecessary prolonged antibiotic use, reduce hospital costs and prevent the further propagation of resistant microbes.

Antibiotic detail: cephalosporins or aminoglycoside + metronidazole or clindamycin and the alternative for allergies being aminoglycoside/ sulbactam or fluoroquinolone

Looking at the same drugs and doses the variable is the timeframe of the medication

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years old
* Negative urine culture within 1 month prior to procedure
* Renal Calculi which would optimally require PCNL for treatment.

Exclusion Criteria:

* Patients <18 years old.
* Patients who are not able to give consent for study
* Patients currently on antibiotics immediately prior to the procedure
* Previous history of sepsis or SIRS from stone manipulations
* Foley catheter in place for greater than 1 week duration
* Patients under going planned, multi-staged procedures
* Immunosuppressed patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2014-09; Primary Completion 2018-03 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zeph Okeke, MD, Principal Investigator — Northwell Health
Locations (2):
- United States (2):
  - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York

REFERENCES:
- [Derived] Griffiths L, Aro T, Samson P, Derisavifard S, Gaines J, Alaiev D, Mullen G, Rai A, Williams T, Patel V, Guanay G, Leavitt D, Hartman C, Smith A, Hoenig D, Okeke Z. Prospective Randomized Trial of Antibiotic Prophylaxis Duration for Percutaneous Nephrolithotomy in Low-Risk Patients. J Endourol. 2023 Oct;37(10):1075-1080. doi: 10.1089/end.2022.0678. PMID 37578113

RESULTS

PARTICIPANT FLOW:
Groups:
- Antibiotics for a 24 Hour Period: Antibiotics for a 24 hour period
  Intervention drug to be determined based on patient history etc.
  cephalosporins: Looking at the same drugs and doses the variable is the timeframe of the medication
  aminoglycoside
  metronidazole
  Clindamycin
  aminoglycoside/ sulbactam: If allergies to above medicines
  Fluoroquinolones
- Continued Antibiotics: Continued antibiotics until the removal of any external catheters
  Intervention drug to be determined based on patient history etc.
  cephalosporins: Looking at the same drugs and doses the variable is the timeframe of the medication
  aminoglycoside
  metronidazole
  Clindamycin
  aminoglycoside/ sulbactam: If allergies to above medicines
  Fluoroquinolones
Period: Overall Study
Arm/Group | Antibiotics for a 24 Hour Period | Continued Antibiotics
Started | 49 | 49
Completed | 49 | 49
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients were randomly assigned to the interventional arm or the control arm through stratified randomization. In addition to perioperative antibiotics, those in the interventional arm only received antibiotic course for up to 24 hours after procedure, while those in the control arm received antibiotics until external catheters were removed based on surgeon preference.
Groups:
- Total: Total of all reporting groups
Arm/Group | Antibiotics for a 24 Hour Period | Continued Antibiotics | Total
Number analyzed (Participants) | 49 | 49 | 98
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 37 | 31 | 68
  >=65 years | 12 | 18 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.1 (11.3) | 59.7 (11.9) | 58.9 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 36 | 36 | 72
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 49 | 49 | 98

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Infectious Complications
Description: Compare the rate of infectious complications following a single-dose of peri-operative protocol (antibiotics for 24 hours as recommended by the American Urological Association Guidelines) with a short-course protocol (antibiotics continued until any external catheters such as nephrostomy tubes are removed) following percutaneous nephrolithotomy. Complication rate differences, primarily infectious complications such as fever, sepsis, systemic inflammatory response.
Time Frame: 0-30 days post-operatively
Population: Patients were randomly assigned to the interventional arm or the control arm through stratified randomization. In addition to perioperative antibiotics, those in the interventional arm only received antibiotic course for up to 24 hours after procedure while those in the control arm received antibiotics until external catheters were removed based on surgeon preference
Measure: Count of Participants; unit: Participants
Arm/Group | Antibiotics for a 24 Hour Period | Continued Antibiotics
Number analyzed (Participants) | 49 | 49
Participants
  Fever | 6 | 7
  SIRS | 6 | 8
  Bacteriuria | 1 | 2
  Bacteremia | 1 | 1

2. Secondary Outcome: Length of Stay (Days)
Description: Length of Hospital Stay After Surgery (days)
Time Frame: 0-30 days post operatively
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Antibiotics for a 24 Hour Period | Continued Antibiotics
Number analyzed (Participants) | 49 | 49
Days | 1.7 (0.8) | 1.5 (1.9)

3. Secondary Outcome: Number of Participants With Associated Clavien Grade of Adverse Event
Description: Overall complication rates are reported based on Clavien-Dindo scale. The numbers reported are recorded Clavien complications. There is only one Clavien complication per patient as such a recorded number indicates one complication of this classification and also one patient with this complication. For example, if a Clavien III is recorded, it is indicating that one patient in that study group had one Clavien III complication.
  Grade I are any deviation from the normal post-operative course not requiring surgical, endoscopic or radiological intervention.
  Grade II complications require drug treatments other than those allowed for Grade I complications; Grade III complications require surgical, endoscopic or radiological intervention either IIIa, not under general anesthesia or IIIb, under general anesthesia. Grade IV are Life-threatening complications. Grade V are most severe and result in death of the patient.
Time Frame: 0 to 30 days after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Antibiotics for a 24 Hour Period | Continued Antibiotics
Number analyzed (Participants) | 49 | 49
Participants
  Grade I | 4 | 3
  Grade II | 2 | 5
  Grade IIIA | 3 | 2
  Grade IIIB | 1 | 2

ADVERSE EVENTS:
Time Frame: All adverse events occurring within the first 30 post-operative days were recorded for each patient.
Description: The primary outcome was the rate of postoperative sepsis further stratified by presence of body temperature >38 degrees Celsius, positive SIRS criteria, bacteremia, or bacteriuria. Adverse events are graded according to Clavien dindo scale, I-V with increasing severity up to V, which is patient death. Serious adverse events are defined by Clavien IIIb or higher, which is defined as requiring an additional procedure with general anesthesia.
Arm/Group | Antibiotics for a 24 Hour Period | Continued Antibiotics
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/49
Serious Adverse Events (participants affected / at risk) | 1/49 | 2/49
Other Adverse Events (participants affected / at risk) | 9/49 | 10/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Antibiotics for a 24 Hour Period (N=49) | Continued Antibiotics (N=49)
Hemothorax/Pneumothorax (Surgical and medical procedures) | 1 (1) | 1 (1) — Puncture of diaphragm during procedure leading to blood or air filling pleural space. This requires patient to have a chest tube placement.
Fevers with Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1) — Post surgical fever with associated hydronephrosis indicates blockage of upper tracts requiring drainage with ureteral stent
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Antibiotics for a 24 Hour Period (N=49) | Continued Antibiotics (N=49)
fevers post operative (Blood and lymphatic system disorders) | 2 (2) | 5 (5) — readmitted for fevers requiring additional antibiotic treatment.
Post operative urinary retention (Renal and urinary disorders) | 3 (3) | 1 (1) — Urinary retention requiring foley catheter placement
Post operative pain (General disorders) | 1 (1) | 1 (1) — return to emergency room for post operative flank pain, resolved with conservative management.
Post operative anemia requiring transfusion (Surgical and medical procedures) | 0 (0) | 1 (1) — Post operative bleeding requiring transfusion
Post-operative embolization (Surgical and medical procedures) | 3 (3) | 2 (2) — post operative delayed bleeding requiring embolization

LIMITATIONS AND CAVEATS:
Procedure included tubeless procedures. While this may aid in generalizability, an element of antibiotic duration variation is unavoidably introduced in this treatment arm. The original design was to have 290 participants, due to the low number of recruitment, this number was reduced to a goal of 100 total with 50 randomized to each arm. This limits the analysis, but ultimately desired measures were achieved.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-18): https://cdn.clinicaltrials.gov/large-docs/61/NCT02579161/Prot_SAP_000.pdf